CLINICAL TRIAL: NCT04180774
Title: An Open-label Study of the Safety and Efficacy of Tag-7 Gene-modified Tumor Cell-based Vaccine in Patients With Locally Advanced or Metastatic Malignant Melanoma or Renal Cell Cancer
Brief Title: Safety and Efficacy of Tag-7 Gene-modified Vaccine in Locally Advanced or Metastatic Malignant Melanoma or Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Collaborators: Institute of Gene Biology Russian Academy of Sciences (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-Ген-М
Record Dates: First submitted 2019-11-22; First posted 2019-11-29 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-11

CONDITIONS: Melanoma; Kidney Cancer
Keywords: gene modified vaccine; tag-7; immunotherapy; tumor cells-based vaccine
MeSH Terms: conditions — Melanoma; Kidney Neoplasms

STUDY DESIGN:
Intervention Model Description: Studied therapy - tag-7 gene-modified vaccine (GMV) is administered intradermally at three spots (3 cm from each other) in the paravertebral area 4-6 weeks after surgery in an adjuvant or metastatic setting in patients with melanoma or kidney cancer (4 cohorts in parallel). Treatment with GMV will be administered as described until the patient experiences either unacceptable toxicity or unequivocal disease progression (PD). Biomarkers were assessed at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Melanoma Adjuvant (Experimental): Patients with completely resected stage III or IV melanoma receiving GMV in the adjuvant setting
  Interventions: Biological: Tag-7 gene modified inactivated tumor cells
- Melanoma Therapeutic (Experimental): Patients with incompletely resected stage III or IV melanoma receiving GMV in the therapeutic setting
  Interventions: Biological: Tag-7 gene modified inactivated tumor cells
- Renal Cell Adjuvant (Experimental): Patients with completely resected stage III or IV kidney cancer receiving GMV in the adjuvant setting
  Interventions: Biological: Tag-7 gene modified inactivated tumor cells
- Renal Cell Therapeutic (Experimental): Patients with incompletely resected stage III or IV kidney cancer receiving GMV in the therapeutic setting
  Interventions: Biological: Tag-7 gene modified inactivated tumor cells

INTERVENTIONS:
Biological: Tag-7 gene modified inactivated tumor cells — Patients received GMV once in three weeks subcutaneously in three points in the paravertebral region. One dose consisted of 10 million transfected and inactivated tumor cells. No dose reduction was allowed.

SUMMARY:
This study was designed to assess the safety and efficacy of inactivated tumor cells genetically modified with the TAG-7 gene as immunotherapy for cancer. Patients with melanoma or kidney cancer were included since they have immune-dependent tumors. Treatment was done in the adjuvant setting after complete cytoreduction of locally advanced or metastatic disease or in the therapeutic setting in patients where complete cytoreduction was impossible.

DETAILED DESCRIPTION:
During the last decade, novel approaches for cancer treatment have been developed. Antitumor vaccines are one of the most promising approaches in tumor immunotherapy. Tumor cells possess low immunogenicity properties due to a number of the not completely understood mechanisms of resistance. One of the ways to overcome it is immune genes transfection. Genes encoding granulocyte-macrophage colony-stimulating factor (GM-CSF), interleukin (IL)-2 and IL-12 have been used most commonly, both in preclinical studies and clinical trials. These cytokines are well known to participate in the systemic immune response. Several studies have shown that the professional antigen-presenting cells (APCs) of the host, rather than the vaccinating tumor cells themselves, are responsible for priming CD4+ and CD8+ T cells, both of which are required to generate systemic antitumor immunity. Recent findings indicate that the adaptive arm of immunity is governed by the innate immune mechanisms that control the co-stimulatory signaling of APCs. Recently, investigators identified a novel gene, tag7, also know as PGRP-S. The insect ortholog of the tag7/PGRP-S was shown to be involved in the innate immune response in Drosophila. In preclinical studies, tag7-modified mouse tumor cells induced a long-lasting T-cell dependent immune response in mice. The effectiveness of antitumor vaccination was demonstrated on different models of mouse tumors, particularly for melanoma cells (M3, B16, F10). Clinically important results of vaccine therapy were achieved in patients with melanoma and renal carcinoma in a number of studies. The results with this treatment are comparable to chemotherapy and immunotherapy. Investigators assume that one has to activate the innate component of immunity first, followed by the activation of the adaptive one, to make anticancer vaccines more effective. Thus, a phase I/II clinical trial has been performed to evaluate the feasibility and toxicity of treatment with autologous tumor cells modified with the tag7 gene, which has been shown to be involved in innate immunity mechanisms,

ELIGIBILITY:
Inclusion Criteria:

1. Signed inform consent form.
2. Patients age ≥ 18 years of age at the time of informed consent.
3. Ability to provide and understand written informed consent prior to any study procedures.
4. Histologically confirmed locally advanced or metastatic MM or RCC.
5. Tumor cell culture should be obtained and successfully transfected before inclusion.
6. No evaluable therapy with a proved survival advantage in the current patient setting.
7. The life expectancy of > 3 months as estimated by the investigator
8. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 -2 at Screening.

Exclusion Criteria:

1. Patient with any out-of-range laboratory values defined as:

   * Serum creatinine > 1.5 × upper limit of normal (ULN) and/or creatinine clearance (calculated using Cockcroft-Gault formula, or measured) < 50 mL/minute
   * Total bilirubin > 2.5 × ULN, except for patients with Gilbert's syndrome who are excluded if total bilirubin > 3.0 × ULN or direct bilirubin > 1.5 × ULN
   * Alanine aminotransferase > 2.5 × ULN
   * Aspartate aminotransferase > 2.5 × ULN
   * Absolute neutrophil count < 1.5 × 109/L
   * Platelet count < 100 × 109/L
   * Hemoglobin < 80 g/L (blood transfusions permitted)
2. History of severe hypersensitivity reactions (eg, anaphylaxis) to other biologic drugs or monoclonal antibodies
3. Any clinically significant unstable disease
4. Presence of symptomatic or untreated central nervous system (CNS) metastases
5. Active infection requiring systemic antibiotic therapy. Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of study drug
6. Known history of human immunodeficiency virus infection (HIV). Testing for HIV status is not necessary unless clinically indicated
7. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection per institutional protocol. Testing for HBV or HCV status is not necessary unless clinically indicated or the patient has a history of HBV or HCV infection
8. Malignant disease, other than that being treated in this study
9. Patients receiving systemic steroid therapy or any other systemic immunosuppressive medication at any dose level, as these may interfere with the mechanism of action of study treatment. Local steroid therapies (eg, otic, ophthalmic, intra-articular or inhaled medications) are acceptable
10. Pregnant, likely to become pregnant, or lactating women (where pregnancy is defined as the state of a female after conception and until the termination of gestation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2001-01-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events rate | From the fist injection to 3 month after the last injection
  CTC AE v.3 was used for safety assesment

SECONDARY OUTCOMES:
Response rate | every 8 weeks until disease progression or therapy completion, then every 3 month for 2 years, every 6 month for the next 2 years and annually thereafter
  To assess the objective response rate (OR) RECIST v1.1 and irRC were used at the final assesment
Concentration of MICA in patient's cultures supernatants | Samples obtained before therapy start
  Factor production by culture of patient's tumor cells, used for vaccine preparation
Concentration of TGF-β1 in patient's cultures supernatants | Samples obtained before therapy start
  Factor production by culture of patient's tumor cells, used for vaccine preparation
Concentration of IL-10 in patient's cultures supernatants | Samples obtained before therapy start
  Factor production by culture of patient's tumor cells, used for vaccine preparation
Concentration of VEGF in patient's cultures supernatants | Samples obtained before therapy start
  Factor production by culture of patient's tumor cells, used for vaccine preparation
Number of T-cells in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) of CD3+ cells in peripheral blood
Number of T-helper lympocytes in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) concentration of CD4+ cells in peripheral blood
Number of Cytotoxic lymphocytes in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) concentration of CD8+ cells in peripheral blood
Number of NK-lymphocytes in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) concentration of CD16+CD56+ cells in peripheral blood
Number of CD38+ cells in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) concentration of CD38+ cells in peripheral blood
Number of HLA-DR+ cells in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) concentration of HLA-DR+ cells in peripheral blood
Number of CD71+ cells in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) concentration of CD71+ cells in peripheral blood
Number of B-lymphocytes cells in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) concentration of CD71+ cells in peripheral blood
Number of CD25+ cells in peripheral blood of patients | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Absolute (10^9/L) concentration of CD25+ cells in peripheral blood
IgA level | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  IgA (g/L) level in serum
IgG level | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  IgG (g/L) level in serum
IgM level | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  IgM (g/L) level in serum
Spontaneous lymphocytes migration | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Lymphocytes migration (U) without stimulation
Kon-A stimulated migration | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Lymphocyte migration after in vitro stimulation with Kon A (% inhibition of migration)
PGA stimulated migration | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Lymphocyte migration after in vitro stimulation with PGA (% inhibition of migration)
Ingestion rate of monocytes | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Ingestion rate (%)
Ingestion rate of neutrophils | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Ingestion rate (%)
Circulating immune complex level | 1-5 days before each therapy cycle during course of therapy (cycle 21 days) through therapy completion, an average of 6 cycles (18 weeks)
  Immune complexes (U) in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Georgy P Georgiev, Study Director — Institute of Gene Biology of the Russian Academy of Sciences
Locations (1):
- N.N. Petrov Research Institute of Oncology Chemotherapy and Innovative Technologies Department, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No